CLINICAL TRIAL: NCT05408754
Title: PARALELL - Pulsed Field Ablation and Pulsed Field CRyoAbLation in PErsistent AtriaL FibrilLation
Brief Title: Pulsed Field Ablation and Pulsed Field CRyoAbLation in PErsistent AtriaL FibrilLation
Acronym: PARALELL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adagio Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-169
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: Pulsed Field Ablation; Pulsed Field CryoAblation; Persistent AF; PFA; PFCA; AF; Adagio Medical
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Field Ablation (PFA) group (Experimental): PsAF patients treated by PFA
  Interventions: Device: Atrial ablation for subject scheduled for a de novo endocardial ablation of symptomatic, drug-refractory PsAF.
- Pulsed Field CryoAblation (PFCA) group (Experimental): PsAF patients treated by PFCA
  Interventions: Device: Atrial ablation for subject scheduled for a de novo endocardial ablation of symptomatic, drug-refractory PsAF.

INTERVENTIONS:
Device: Atrial ablation for subject scheduled for a de novo endocardial ablation of symptomatic, drug-refractory PsAF. — Treatment will include the isolation of pulmonary veins (PVIs), and isolation of the left atrial posterior wall (PWI). A right atrial cavo-tricuspid line for bi-directional block may be performed at discretion and clinical judgment of the investigator

SUMMARY:
A prospective, two-arm, multi-center, randomized, open-label, pre-market, First-in-Human clinical study designed to provide safety and performance data regarding the use of the Adagio PFA and PFCA Systems in the treatment of PsAF.

DETAILED DESCRIPTION:
Enrolled subjects will be treated (ablation) with the Adagio PFA or PFCA System in a 1:1 randomized fashion.

Treatment will include the isolation of pulmonary veins (PVIs), and isolation of the left atrial posterior wall (PWI), and CTI at the discretion and clinical judgment of the investigator.

Data will be collected throughout 12-month follow up period to assess safety and performance of the device. Recurrence of atrial arrhythmias is measured by 12-lead ECGs and 48-hour continuous ECG recording (Holter).

ELIGIBILITY:
Inclusion Criteria:

IC 1 Male or female between the ages of 18 - 80 years

IC 2 Currently scheduled for an ablation of symptomatic persistent (> 7 days) atrial fibrillation within the past year documented by ECG or Continuous Holter monitoring

IC 3 Refractory to at least one class I or III AAD. (Refractory defined as not effective or not tolerated)

IC 4 Willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full length of the study

IC 5 Willingness and ability to give an informed consent

Exclusion Criteria:

EC 1 In the opinion of the Investigator, any known contraindication to an atrial ablation, TEE, or anticoagulation. Including but not limited to the identification of any atrial thrombus or evidence of sepsis

EC 2 Continuous AF lasting longer than 12-months

EC 3 History of previous left atrial ablation or surgical treatment for AF/AFL/AT

EC 4 AF secondary to electrolyte imbalance, active thyroid disease, or any other reversible or non-cardiac cause

EC 5 Structural heart disease as described below:

1. Left ventricular ejection fraction (LVEF) < 40% based on most recent TTE
2. Left atrial size > 55 mm (parasternal long axis view) documented within 6-months of screening
3. NYHA Class III or IV heart failure documented within the previous 12-months
4. An implanted pacemaker or ICD
5. Previous cardiac surgery, ventriculotomy, or atriotomy (excluding atriotomy for CABG),
6. Previous cardiac valvular surgical or percutaneous procedure, or prosthetic valve
7. Interatrial baffle, closure device, patch, or PFO occluder
8. Presence of a left atrial appendage occlusion device
9. Presence of any pulmonary vein stenting devices
10. Coronary artery bypass graft (CABG) or PTCA procedure within six (6) months prior to procedure
11. Unstable angina or ongoing myocardial ischemia
12. Myocardial infarction within the previous six (6) months prior to procedure
13. Moderate or severe mitral insufficiency or stenosis based on most recent TTE
14. Atrial myxoma
15. Significant congenital anomaly

EC 6 BMI > 40

EC 7 Any previous history of cryoglobulinemia (for those patients randomized to the PFCA arm)

EC 8 History of blood clotting or bleeding disease

EC 9 History of severe COPD requiring steroid use in the previous 12-months

EC 10 History of severe sleep apnea (AHI > 30) not currently treated with a CPAP machine or other mechanical device

EC 11 Stroke or TIA within the last year.

EC 12 Any prior history or current evidence of hemidiaphragmatic paralysis

EC 13 Pregnant or lactating (current or anticipated during study follow-up

EC 14 Current enrollment in any other study protocol where testing or results from that study may interfere with the procedure or outcome measurements for this study

EC 15 Any other conditions such as, mental illness, addictive disease, terminal illness with a life expectancy of less than two years, extensive travel away from the research center that may lead to non-compliance with the protocol procedure or follow up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint for Safety | Up to 7 days following the ablation procedure
  Analysis of the proportion of subjects who are free from device/procedure-related Major Adverse Events that occur during or following the ablation procedure
Primary Procedural Performance Outcome | Procedure
  Analysis of the evidence of procedural electrical isolation of all pulmonary veins, posterior wall, and bidirectional block (if applicable) across all other ablation lines using the study device.

SECONDARY OUTCOMES:
One-Year Safety | 12 months
  Recording and analysis of all identified serious adverse events and serious adverse device effects through 12 months post-procedure.
One-Year Performance | 12 months
  Proportion of subjects receiving a single ablation procedure who has freedom from any documented left atrial arrhythmia (AF/AFL/AT) lasting longer than 30 seconds following the Blanking Period (3-months ± 14-days post index ablation) using a continuous 48-hour ECG recording through 12 months post-procedure.
Procedural Performance - ablation time | procedure
  Ablation time defined as the total time for energy delivery to achieve PVI, PWI, and CTI (if applicable)
Procedural Performance - procedure time | procedure
  Total procedure time defined as the time from first venous access to the removal of the catheters from the heart at the end of the procedure
Procedural Performance - fluoroscopy time | procedure
  Procedure fluoroscopy time
Procedural Performance - intraprocedural PV reconnection rate | procedure
  The rate of intraprocedural PV reconnection - defined as confirmed conduction across a PVI line during the 20-minute waiting period to confirm PVI
Procedural Performance - AAD use | procedure and up to 12-month
  Recording of the use of AADs in the follow up period beyond a 90-day blanking period
Procedural Performance - repeat ablation | procedure and up to 12-month
  Number of repeat ablations within and following the blanking period

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Principal Investigator — McGill University Health Centre; Montreal, Canada
Locations (6):
- Onze-Lieve-Vrouwziekenhuis (OLV), Aalst, Belgium
- McGill University Health Centre (MUHC), Montreal General Hospital (MGH), Montreal, Quebec, Canada
- Nemocnice Na Homolce, Prague, Czechia
- Blackrock Health, Dublin, Ireland
- St Antonius Ziekenhuis, Nieuwegein, Netherlands
- St George'S University Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No